CLINICAL TRIAL: NCT03317288
Title: Effect of Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in People With Spinal Cord Injury
Brief Title: Alternating Pressure Overlay on Weight Bearing Tissue Tolerance in People With Spinal Cord Injury
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Collaborators: Dabir Surfaces Inc (Industry)
Responsible Party: Principal Investigator, Yi-Ting Tzen, Assistant professor, University of Illinois at Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017-0215
Record Dates: First submitted 2017-10-10; First posted 2017-10-23 (Actual); Results first posted 2021-06-09 (Actual); Last update posted 2021-06-09 (Actual); Status verified 2021-05

CONDITIONS: Spinal Cord Injuries; Pressure Ulcer
Keywords: spinal cord injury; pressure ulcer; laser Doppler flowmetry
MeSH Terms: conditions — Spinal Cord Injuries; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: Repeated measures design. Subject serves as his or her own control.
Masking Description: Here is no masking of the intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- SCI subjects (Other): The subject act as his or her own control. Each subject will undergo two procedures, intervention: alternating pressure overlay on top of standard operation room overlay, vs. control: operation room overlay.
  Interventions: Device: Dabir Air overlay

INTERVENTIONS:
Device: Dabir Air overlay — The Dabir Air overlay is a low profile alternating pressure overlay that is designed to place on top of mattress and operation room table.

SUMMARY:
The purpose of this study is to test if the newly-developed Dabir alternating pressure (AP) overlay could be beneficial to preventing skin damage during daily activities, such as lying in bed. Specifically, the study is being done to test if the Dabir AP overlay could be used to increase skin tolerance when lying in bed for an extended period of time (40 minutes), including reducing pressure and increasing skin blood flow (amount of blood supply to oxygen and nutrients to skin) as compared to regular operation room (OR) overlay.

A total of 20 participants with spinal cord injury will be recruited. Subjects will undergo study procedures including: AP and Control protocols. Skin blood flow and interface pressure will be collected non-invasively (from outside the body) during both protocols. During AP protocols, subject will be asked to lie on side (10 min), on back on AP overlay (40 min), on side (30 min), on back on OR overlay (40 min), and on side (10 min). During Control protocol, subject will be asked to lie on side (10 min), on back on OR overlay (40 min), and on side (10 min). Subject will then proceed to vascular control measures, including: non-invasive skin blood flow and tissue oxygen measurements with mild heating and electrical stimulation. Findings from this study will help us understand the effectiveness of the AP overlay on skin blood flow response during prolonged lying in bed.

DETAILED DESCRIPTION:
Tissue ischemia is one of the main etiologies of pressure injury. It is inevitable during bed-ridden and wheelchair bound conditions, such as spinal cord injury (SCI), or prolonged surgery procedure in the operating room. Active alternating pressure (AP) mattresses are covered by Medicare policy for patients with multiple/large stage 2/ stage 3 pressure injuries to relief interface pressure and prevent recurrence of pressure injuries. Previous studies demonstrated that the protective mechanisms of AP on pressure injury include redistribution of surface pressure, and allowing more blood supplies while lying on the support surface. The Dabir AP overlay is low profile yet possesses similar characteristics as other AP mattresses on the market; it is intended for clinical use, such as operation room (OR) where AP mattresses may not be an option. We expect Dabir AP overlay will be beneficial to people at risk of pressure injury by maintaining the blood supply during weight bearing condition.

The objective of this study is to evaluate the protective mechanisms of Dabir AP overlay on weight bearing tissue of people with chronic spinal cord injury (SCI). Our central hypothesis is that the Dabir AP overlay will cause lower amount of interface pressure and allow more skin blood flow during weight bearing as compared to regular OR overlay.

Each subject will undergo two study protocols: AP and control, and the order of the protocols will be randomized by drawing one envelope from the envelope pool. We will start with a pool of total 20 envelopes (10 envelopes indicating AP protocol first, and 10 envelopes indicating control protocol first). A 30-minute washout period will be provided in between the two protocols. Two Laser Doppler flowmetry (LDF) flat probes (moor instrument, Wilmington, DE) will be taped to the sacrum and one heel to collect the skin blood flow response throughout both AP and control protocols. A whole body pressure mapping system will be used between the subject and the overlay to collect the inter pressure data. For the AP cycle, we will use four 10-minute cycles (5 minutes of high pressure and 5 minutes of low pressure).

AP protocol: The subject will first lie on his/her side quietly for 10 minutes to collect the baseline skin blood flow, followed by lying supine on the Dabir AP overlay for 40 minutes, and then side lying for 30 minutes to collect the first reactive hyperemic response. To test the effect of preconditioning, the subject will then lie supine on the OR overlay for 40 minutes followed by side lying for 30 minutes for the second reactive hyperemic response.

Control protocol: The subject will first lie on his/her side quietly for 10 minutes to collect the baseline skin blood flow, followed by lying supine on the OR overlay for 40 minutes, and then side lying for 30 minutes to collect the reactive hyperemic response for control protocol.

The PI, or key personnel will then collect the vascular control measures, including the heat hyperemic (HH) blood flow response, and the skin vasomotor response. A non-invasive combined laser Doppler and white light reflectance spectroscopy (LDF-WLRS) probe (CP2T-1000, Moor Instrument, Wilmington, DE) will be used for both measures.

HH blood flow response will be measured at the sacrum and one heel while the subject is in side-lying position. HH will be induced with the heater at the tip of the probe head (41°C for 5 minutes). This HH measure will take approximately 7 minutes (2 min-baseline, 5 min-heating) per location. In total, the HH measures will take up to 15 minutes to complete.

The skin vasomotor response will be induced using cutaneous electrical stimulation (3-10 mA, 0.2-1.0 ms pulses at 20 Hz, 1 s trains) delivered via 1 cm Ag-AgCl surface electrodes applied bilaterally (4 cm apart) to the forehead (above lesion) and the abdominal wall (below lesion) while the subject is in a semi-reclined position.12 For each site, 5-8 stimuli will be delivered randomly. CP2T-1000 probe will be used to collect SBF and tissue oxygenation data at pulp of the second finger and toe. Subject will be in a semi-reclined position (about 30° from horizontal plane) during this protocol, and it will take up to 15 minutes to complete this protocol.

Pressure mapping of wheelchair: (approximately 10 minutes) The subject will be asked to transfer back to his/her wheelchair with the pressure mapping system placed between the wheelchair and the subject to collect the interface pressure data. The pressure mapping system is the same as that used between the subject and overlay to collect the interface pressure data.

ELIGIBILITY:
Inclusion Criteria:

* have had spinal cord injury for more than one year
* have injury level at T10 or above
* not ambulatory and use a wheelchair for mobility
* none smokers or able to refrain from smoking four hours prior to and during the study

Exclusion Criteria:

* current pressure ulcer
* history of diabetes mellitus
* history of cardiovascular diseases
* history of hypertension
* history of pulmonary diseases
* pregnant women (based on a positive pregnancy test)
* Non-English speakers

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2019-03-31 (Actual); Study Completion 2019-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Yi-Ting Tzen, PhD, Principal Investigator — Assistant Professor
Locations (1):
- University of Illinois at Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | SCI Subjects
Started | 15
Completed | 15
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | SCI Subjects
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 41.87 (14.89)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: African American | 11
  Ethnicity: Asian | 1
  Ethnicity: Caucasian | 1
  Ethnicity: Hispanic | 2
Region of Enrollment [Number; unit: participants]
  United States | 15
body mass index [Mean (Standard Deviation); unit: kg/m2] | 26.81 (4.13)
duration of spinal cord injury [Mean (Standard Deviation); unit: years] | 17 (14.62)
level of spinal cord injury [Count of Participants; unit: Participants]
  At T6 and above | 6
  Below T6 | 9
American Spinal Injury Association Scale score [Count of Participants; unit: Participants]
  Complete | 5
  Incomplete | 10

OUTCOME MEASURES:

1. Primary Outcome: Sacral Skin Blood Flow During Supine Lying
Description: Sacral skin blood flow measured using laser Doppler flowmetry system (moor instrument) during supine lying on operating room pad with and without alternating pressure overlay
Time Frame: 40 minutes, the inflation-deflation cycle alternates every 10 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: arbitrary unit
Groups:
- Alternating Pressure -- Inflation Cycle: Averaged skin blood flow during the inflation cycle of the alternating pressure
- Alternating Pressure -- Deflation Cycle: Averaged skin blood flow during the deflation cycle of the alternating pressure
- Control (Operating Room Pad Only): Averaged skin blood flow during supine lying on the operating room pad only (without alternating pressure overlay)
Arm/Group | Alternating Pressure -- Inflation Cycle | Alternating Pressure -- Deflation Cycle | Control (Operating Room Pad Only)
Number analyzed (Participants) | 15 | 15 | 15
arbitrary unit | 12.65 (12.45) | 15.54 (15.33) | 11.96 (10.26)

2. Primary Outcome: Heel Skin Blood Flow During Supine Lying
Description: Heel skin blood flow measured using laser Doppler flowmetry system (moor instrument) during supine lying on operating room pad with and without alternating pressure overlay
Time Frame: 40 minutes, the inflation-deflation cycle alternates every 10 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Alternating Pressure -- Inflation Cycle | Alternating Pressure -- Deflation Cycle | Control (Operating Room Pad Only)
Number analyzed (Participants) | 15 | 15 | 15
arbitrary unit | 15.10 (20.78) | 27.92 (32.15) | 10.43 (11.16)

3. Primary Outcome: Sacral Peak Interface Pressure During Supine Lying
Description: Sacral peak interface pressure measured using pressure mapping system during supine lying on operating room pad with and without alternating pressure overlay. This is the maximum interface pressure of the nine pressure cells located at the sacrum.
Time Frame: 40 minutes, the inflation-deflation cycle alternates every 10 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Alternating Pressure -- Inflation Cycle: Averaged peak interface pressure during the inflation cycle of the alternating pressure
- Alternating Pressure -- Deflation Cycle: Averaged peak interface pressure during the deflation cycle of the alternating pressure
- Control (Operating Room Pad Only): Averaged peak interface pressure during supine lying on the operating room pad only (without alternating pressure overlay)
Arm/Group | Alternating Pressure -- Inflation Cycle | Alternating Pressure -- Deflation Cycle | Control (Operating Room Pad Only)
Number analyzed (Participants) | 15 | 15 | 15
mmHg | 89.27 (53.92) | 51.47 (30.18) | 114.13 (60.97)

4. Primary Outcome: Sacral Averaged Interface Pressure During Supine Lying
Description: Sacral averaged interface pressure measured using pressure mapping system during supine lying on operating room pad with and without alternating pressure overlay. This is the averaged interface pressure of the nine pressure cells located at the sacrum.
Time Frame: 40 minutes, the inflation-deflation cycle alternates every 10 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Alternating Pressure -- Inflation Cycle: Averaged interface pressure during the inflation cycle of the alternating pressure
- Alternating Pressure -- Deflation Cycle: Averaged interface pressure during the deflation cycle of the alternating pressure
- Control (Operating Room Pad Only): Averaged interface pressure during supine lying on the operating room pad only (without alternating pressure overlay)
Arm/Group | Alternating Pressure -- Inflation Cycle | Alternating Pressure -- Deflation Cycle | Control (Operating Room Pad Only)
Number analyzed (Participants) | 15 | 15 | 15
mmHg | 57.21 (28.54) | 36.16 (18.47) | 81.50 (46.39)

5. Primary Outcome: Heel Peak Interface Pressure During Supine Lying
Description: Heel peak interface pressure measured using pressure mapping system during supine lying on operating room pad with and without alternating pressure overlay. This is the maximum interface pressure of the nine pressure cells located at the heel.
Time Frame: 40 minutes, the inflation-deflation cycle alternates every 10 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Alternating Pressure -- Inflation Cycle | Alternating Pressure -- Deflation Cycle | Control (Operating Room Pad Only)
Number analyzed (Participants) | 15 | 15 | 15
mmHg | 52.49 (21.21) | 26.79 (12.91) | 53.05 (18.22)

6. Primary Outcome: Heel Averaged Interface Pressure During Supine Lying
Description: Heel averaged interface pressure measured using pressure mapping system during supine lying on operating room pad with and without alternating pressure overlay. This is the averaged interface pressure of the nine pressure cells located at the heel.
Time Frame: 40 minutes, the inflation-deflation cycle alternates every 10 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Alternating Pressure -- Inflation Cycle | Alternating Pressure -- Deflation Cycle | Control (Operating Room Pad Only)
Number analyzed (Participants) | 15 | 15 | 15
mmHg | 37.88 (17.27) | 14.60 (8.37) | 34.83 (16.62)

7. Secondary Outcome: Post Alternating Pressure Sacral Skin Blood Flow
Description: Sacral skin blood flow measured using laser Doppler flowmetry system (moor instrument) during supine lying on operating room pad after 40 minutes on operating room pad with or without alternating pressure and a 30 minutes washout period.
Time Frame: 40 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: arbitrary unit
Groups:
- Post Alternating Pressure: Averaged skin blood flow during supine lying after lying on operating room pad with alternating pressure
- Control: Averaged skin blood flow during supine lying after operating room pad only
Arm/Group | Post Alternating Pressure | Control
Number analyzed (Participants) | 15 | 15
arbitrary unit | 15.78 (15.82) | 11.96 (10.26)

8. Secondary Outcome: Post Alternating Pressure Sacral Peak Interface Pressure
Description: Sacral peak interface pressure during supine lying on operating room pad after 40 minutes on operating room pad with or without alternating pressure and a 30 minutes washout period.
Time Frame: 40 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Post Alternating Pressure: Averaged peak interface pressure during supine lying after lying on operating room pad with alternating pressure
- Control: Averaged peak interface pressure during supine lying after operating room pad only
Arm/Group | Post Alternating Pressure | Control
Number analyzed (Participants) | 15 | 15
mmHg | 104.62 (58.17) | 114.13 (60.97)

9. Secondary Outcome: Post Alternating Pressure Sacral Averaged Interface Pressure
Description: Sacral averaged interface pressure during supine lying on operating room pad after 40 minutes on operating room pad with or without alternating pressure and a 30 minutes washout period.
Time Frame: 40 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: mmHg
Groups:
- Post Alternating Pressure: Averaged interface pressure during supine lying after lying on operating room pad with alternating pressure
- Control: Averaged interface pressure during supine lying after operating room pad only
Arm/Group | Post Alternating Pressure | Control
Number analyzed (Participants) | 15 | 15
mmHg | 81.07 (48.62) | 81.50 (46.39)

10. Secondary Outcome: Post Alternating Pressure Heel Skin Blood Flow
Description: Heel skin blood flow measured using laser Doppler flowmetry system (moor instrument) during supine lying on operating room pad after 40 minutes on operating room pad with or without alternating pressure and a 30 minutes washout period.
Time Frame: 40 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: arbitrary unit
Arm/Group | Post Alternating Pressure | Control
Number analyzed (Participants) | 15 | 15
arbitrary unit | 16.31 (29.18) | 10.43 (11.16)

11. Secondary Outcome: Post Alternating Pressure Heel Peak Interface Pressure
Description: Heel peak interface pressure during supine lying on operating room pad after 40 minutes on operating room pad with or without alternating pressure and a 30 minutes washout period.
Time Frame: 40 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Post Alternating Pressure | Control
Number analyzed (Participants) | 15 | 15
mmHg | 47.69 (16.21) | 53.05 (18.22)

12. Secondary Outcome: Post Alternating Pressure Heel Averaged Interface Pressure
Description: Heel averaged interface pressure during supine lying on operating room pad after 40 minutes on operating room pad with or without alternating pressure and a 30 minutes washout period.
Time Frame: 40 minutes
Population: All participants with spinal cord injury. Each participant serves as his/her own control.
Measure: Mean (Standard Deviation); unit: mmHg
Arm/Group | Post Alternating Pressure | Control
Number analyzed (Participants) | 15 | 15
mmHg | 30.35 (17.59) | 34.83 (16.62)

ADVERSE EVENTS:
Time Frame: Total study duration
Description: The reason why the number of participants at risk for serious adverse events and all-cause mortality is zero is because the intervention is an FDA exempt overlay on top of an operating room pad. Lying on top of the overlay pose no risk of mortality or any serious adverse events.
Arm/Group | SCI Subjects
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

LIMITATIONS AND CAVEATS:
Small sample size with very strict criteria, results could not be generalized to other population.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2017-04-04): https://cdn.clinicaltrials.gov/large-docs/88/NCT03317288/Prot_SAP_000.pdf
  • Informed Consent Form (2017-05-08): https://cdn.clinicaltrials.gov/large-docs/88/NCT03317288/ICF_001.pdf